CLINICAL TRIAL: NCT06199700
Title: An Exploratory Trial of Esketamine for the Treatment of Rett Syndrome
Brief Title: Esketamine for the Treatment of Rett Syndrome
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EskRTT2023; XE2023-ETBJ-D01 (Other Grant/Funding Number: Fujian Province Clinical Key Specialty Construction Project)
Record Dates: First submitted 2023-11-21; First posted 2024-01-10 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Rett Syndrome
Keywords: Rett syndrome; Esketamine; efficacy; safety
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Esketamine treatment (Experimental): Esketamine, diluted with 20ml Saline at a dose of 0.25mg/kg, intravenously for 40 minutes, once a week; 5 weeks in total.
  Interventions: Drug: Esketamine hydrochloride

INTERVENTIONS:
Drug: Esketamine hydrochloride — Intravenous infusion of Ketamine

SUMMARY:
The goal of this interventional study is to learn about the efficacy and safety of Esketamine for treating children with Rett syndrome (RTT).

The main questions it aims to answer are:

* whether Esketamine treatment is effective in improving symptom severity for RTT.
* whether Esketamine is safe in the treatment of RTT. Participants will receive a weekly intravenous infusion of Esketamine for five weeks and will be assessed for disease severity and drug safety.

ELIGIBILITY:
Inclusion Criteria:

* Classic/typical RTT
* Causing mutation in MECP2 gene
* Stable pattern of seizures, or has had no seizures at least 8 weeks

Exclusion Criteria:

* Use of other drugs that interact with Esketamine: thyroxine, meglumine diatrizoate, aminophylline, diazepam or midazolam, drugs for antihypertension or central nervous depressants, halogenated general anesthetics (e.g., halothane), tubocurarine, atracurium
* Condition with hypertension, high cerebrospinal fluid pressure, and high intraocular pressure
* Unstable systemic illness other than Rett syndrome: current clinically significant cardiovascular, endocrine (such as hypo- or hyperthyroidism, type 1 diabetes, or uncontrolled type 2 diabetes), renal, hepatic, respiratory, or gastrointestinal disease (such as celiac disease or inflammatory bowel disease), or major surgery planned during the study
* Clinically important variations in medication use

Ages: 5 Years to 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of treatment with Esketamine in girls with RTT | baseline, week 5, and month 6
  Rett Syndrome Behaviour Questionnaire (RSBQ) total score; Minimum value 0; Maximum values 90; higher scores mean a worse outcome.
Incidence of Adverse events | baseline, week 5
  Safety of treatment with Esketamine in girls with RTT
Co-outcome for efficacy of treatment with Esketamine in girls with RTT | baseline, week 5, and month 6
  Clinical Global Impressions Scale-improvement (CGI-I) score; Minimum value 0; Maximum values 7; higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) | baseline, week 5, and month 6
  Total score，; Minimum value 0; Maximum values 28; higher scores mean a worse outcome.
Griffiths Scales of Child Development | baseline, week 5, and month 6
  Development quotient; Minimum value 0; Maximum values 96; higher scores mean a better outcome.
Revised-Motor Behavior Assessment scale (R-MBA) | baseline, week 5, and month 6
  Subscale score, 0-100, higher sores means a worse outcome
Rett Syndrome Severity Scale (RSSS) | baseline, week 5, and month 6
  Subscale score, 0-21, higher sores means a worse outcome
Sleep improvement by Esketamine treatment | baseline, week 5, and month 6
  Sleep record
Behavior observation | baseline, week 5, and month 6
  Unusual hand movements duration per hour
Brain image change | baseline, week 5, and month 6
  Magnetic Resonance Imaging (MRI)；brain network connectivity
Brain function change | baseline, week 5, and month 6
  Electroencephalogram (EEG); brain-wave activity

CONTACTS AND LOCATIONS:
Overall Officials: Huiping Li, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Xiamen Children's Hospital (Children's Hospital of Fudan University at Xiamen), Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: starting 6 months after publication，for one year